CLINICAL TRIAL: NCT04099017
Title: Effectiveness of Mulligan Joint Mobilizations and Trunk Stabilization Exercises Versus Isometric Knee Strengthening in the Management of Knee Osteoarthritis: a Randomized Controlled Trial
Brief Title: Mulligan Manual Therapy and Trunk Stabilization Exercises Versus Isometric Knee Strengthening on Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Shaikh Nabi Bukhsh Nazir, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IPM&R/DUHS-19/
Record Dates: First submitted 2019-09-18; First posted 2019-09-23 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Osteoarthritis, Knee
Keywords: manual therapy; kinesiotape; Excercise therapies; isometric contraction; muscle strength
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: After confirming eligibility, the physiotherapist performing intervention obtained treatment assignment (S.S. Ali). The subject will not be aware of the group allocation and different time slot will be given for the intervention. Another physiotherapist who will not be aware of allocation concealment, record the reading of outcomes at the baseline, after three and six weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mulligan mobilization group (Experimental): This study ARM will received Mulligan joint mobilization and concomitant therapies in this group.
  The following are the brief detail of therapy
  1. Mulligan joint mobilization in Non-weight bearing (NWB):
  2. Knee strengthening
  3. Kinesiotaping
  Interventions: Other: Mulligan Joint mobilization
- Trunk stabilization group (Experimental): This study ARM will received Trunk stabilization exercises and concomitant therapies in this group.
  The following are the brief detail of therapy:
  1. Trunk stabilization i. modified supermen extension exercise ii. Back bridge: iii. Unilateral back bridge:
     Iv. lateral step up:
  2. Knee strengthening i. Isometric quadriceps exercise: ii. Straight leg raising (SLR) exercise:
  3. Kinesiotaping:
  Interventions: Other: Trunk stabilization group
- Knee strengthening group (Other): This study ARM will received Knee strengthening exercises and concomitant therapies in this group.
  The following are the brief detail of therapy:
  1. Knee strengthening i. Isometric quadriceps exercise ii. Straight leg raising (SLR) exercise:
  2. Kinesio-taping:
  Interventions: Other: Knee strengthening group

INTERVENTIONS:
Other: Mulligan Joint mobilization — This study ARM will received Mulligan joint mobilization and concomitant therapies in this group.
  The following are the brief detail of therapy
  1. Mulligan joint mobilization in Non-weight bearing (NWB) to weight-bearing (WB) 6 -10 Reps and 3 sets/ session.
     Procedural detail:
     Joint mobilization will be performed in sagittal, frontal and transverse direction, following glide will be preferred will depend on patient adherence to the joint mobilization. Mobilization will be progress from NWB to WB according to patient compliance 27
  2. Knee strengthening Type of exercise: Knee Isometric Strengthening exercises. Intensity: 10 reps Frequency: At 1st week one set of all knee exercise will be performed then it will be progressed to 2 sets at 3 weeks, and these exercises will be progressed to three sets until the 6 weeks
  3. Kinesiotaping:
  Arms: Mulligan mobilization group
Other: Trunk stabilization group — This study ARM will received Trunk stabilization exercises and concomitant therapies in this group.
  The following are the brief detail of therapy:
  1. Trunk stabilization Area: Trunk Type of exercise: Stabilization exercise Intensity: 6-8 reps Frequency: 3 sets per session and 30 second duration break between sets
     Procedural detail:
     i. modified supermen extension exercise ii. Back bridge: iii. Unilateral back bridge:
     Iv. lateral step up:
  2. Knee strengthening Area: Knee Joint Type of exercise: Knee Isometric Strengthening exercises. Intensity: 10 reps Frequency: At 1st week one set of all knee exercise will be performed then it will be progressed to 2 sets at 3 weeks, and these exercises will be progressed to three sets until the 6 weeks
     Procedural detail:
     i. Isometric quadriceps exercise: ii. Straight leg raising (SLR) exercise:
  3. Kinesiotaping:
  Arms: Trunk stabilization group
Other: Knee strengthening group — This study ARM will received Knee strengthening exercises and concomitant therapies in this group.
  The following are the brief detail of therapy:
  1. Knee strengthening Area: Knee Joint Type of exercise: Knee Isometric Strengthening exercises. Intensity: 10 reps Frequency: At 1st week one set of all knee exercise will be performed then it will be progressed to 2 sets at 3 weeks, and these exercises will be progressed to three sets until the 6 weeks
     Procedural detail:
     i. Isometric quadriceps exercise ii. Straight leg raising (SLR) exercise:
  2. Kinesio-taping:
  Muscle stretch method will be applied which involves one Y and two I straps: The Y-shaped tape base will be affixed over the top of patella then pulls up his/her knee to its maximum bending capacity then both end of Y strip is placed around the patella ending on the tibial tuberosity. Then reinforcing I-tape will be affixed at the origin and insertion of MCL and LCL. Tape will be change in every session.
  Arms: Knee strengthening group

SUMMARY:
Knee joint arthritis posses a serious health problem and caring for an individual with knee osteoarthritis (KOA) produces a great burden on society. Knee joint pain is associated with physical activity while performing various activities of daily living (ADL) in patients with early and severe osteoarthritis (OA). In addition to knee pain, physical function or daily activity is strongly influenced by the severity of Osteoarthritis of the knee. Mulligan joint mobilization with movement provides evident effects on decreasing the pain and restoring the joint biomechanics. Trunk stabilization exercise will improve the stability of trunk which distributes the weight of body evenly on both feets. The aim of this study is to determine the effects of mulligan joint mobilization and trunk stabilization exercise on pain, disability and submaximal exercise performance in KOA.

DETAILED DESCRIPTION:
A randomized control trial will be conducted at IPM&R on 60 subjects with knee osteoarthritis and age between 40-60 years. Initial screening of the subjects will be carried out by the referring consultant. Subjects who fulfilled the study criteria will be recruited using computer generated random sampling after explaining the study objective and taken written informed consent. All participants will be evaluated using visual analogue scale, Knee injury and Osteoarthritis Outcome Score and 6-minute walk test for pain severity, functional limitation and submaximal exercise capacity at 1st, 3rd and 6th week. The subjects will be allocated into three groups through computer generated random allocation. Group 1 will receive mulligan mobilization with kinesiotaping and knee strengthening. Group 2 will receive trunk stabilization exercise, knee strengthening and Kinesiotaping. Group 3 will receive knee strengthening along with kinesiotaping. A drop-out rate of 9 will be taken. Recorded data will be entered and analysed using SPSS version 21. Mean and SD will be calculated of quantitative variables like age, pain, knee related function, submaximal exercise capacity and stair climb by using repeated measure ANOVA. For pair wise comparison, post hoc tukey will be applied. Value of equal to or less than 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* - Both gender (female and male) patients
* Age between 40 - 60
* Knee osteoarthritis Grade I & II on Kellgren and Lawrence (K/L) criteria
* Prediagnosed case of knee OA as per the American College of Rheumatology (ACR).

Exclusion Criteria:

* Known skin allergies
* Sensory-motor dysfunction of lower extremity
* Severe joint deformity of lower extremity
* Post Traumatic Arthritis
* Constitutional Symptoms (Fever, Malaise, Weight Loss and high blood pressure)
* Knee Intraarticular injection in past 3 months
* Acute low back pain
* History of spinal surgery
* Subject using assistive devices for ambulation i.e. cane, walkers, sticks
* Refused to give consent
* Body Mass Index > 30 kg/m2
* Received physiotherapy treatment in the past 3 months
* Visual Analogue Scale <4
* Patellofemoral joint arthritis will be excluded

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-03-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline Knee injury and Osteoarthritis Outcome Score (KOOS) at 6 weeks | baseline and post intervention (week 6 - the analysis will be conducted on the first week immediately after the end of the training
  The Knee injury and Osteoarthritis Outcome Score (KOOS) is a self reported specific joint measure developed to assess a broad spectrum of patients with knee injuries and OA, for pain and other symptoms, function in daily life, function in sports and recreation, and quality of knee-related life, being easy to use, evaluating the short- and long-term health problems related to the knee joint.
  The KOOS contains 42 items covering five subscales: pain, other symptoms, activities of daily living, sport and leisure activities and quality of life. A score of 0 (extreme problems) 100 (smoothly) can be obtained separately for each sub-range.

SECONDARY OUTCOMES:
Visual Analogue Scale | baseline, 3 weeks and 6 weeks
  It measures the subjective of pain ranges from 10-cm lines with defined cut off scores. The correlation between vertical and horizontal orientations of the VAS is 0.99 . Aggregate score ranges for this screening tool starting with 0-10. Scores between 0-4 means mild pain. Scores between 4-7 indicates moderate pain. Scores between 7-10 means severe pain. pain severity will be assessed at rest and during stairs ascending and descending
Knee injury and Osteoarthritis Outcome Score (KOOS) | baseline, 3 weeks and 6 weeks
  The Knee injury and Osteoarthritis Outcome Score (KOOS) is a self reported specific joint measure developed to assess a broad spectrum of patients with knee injuries and OA, for pain and other symptoms, function in daily life, function in sports and recreation, and quality of knee-related life, being easy to use, evaluating the short- and long-term health problems related to the knee joint.
  The KOOS contains 42 items covering five subscales: pain, other symptoms, activities of daily living, sport and leisure activities and quality of life. A score of 0 (extreme problems) 100 (smoothly) can be obtained separately for each sub-range.
6 Minute Walk Test | baseline, 3 weeks and 6 weeks
  The 6-min walk test (6 MWT) is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes. Bright colour tapes will be used to mark the 12m walkway at each end. It will be ensured that the environment will be free from hazards and readings will be recorded by blind assessor. Participant will be instructed to wear comfortable shoes.
Stairs Climb Test | baseline, 3 weeks and 6 weeks
  Stair climb test is used to measure the total time taken by the participant to ascend and descend stair onto with a step length of 16-cm (ICC=0.90). If safety is of concern, the assessor should guard behind the participant going up the stairs and to the side coming down the stairs. If there is no concern for safety, the tester should remain at the start/finish position on the ground landing

CONTACTS AND LOCATIONS:
Overall Officials: SHAIKH NABI B NAZIR, MSAPT, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Dow University of Health Sciences & Institute of Physical Medicine and Rehabilitation, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 3 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Background] Nam CW, Park SI, Yong MS, Kim YM. Effects of the MWM Technique Accompanied by Trunk Stabilization Exercises on Pain and Physical Dysfunctions Caused by Degenerative Osteoarthritis. J Phys Ther Sci. 2013 Sep;25(9):1137-40. doi: 10.1589/jpts.25.1137. Epub 2013 Oct 20. PMID 24259931
- [Derived] Nazir SNB, Rathore FA. Efficacy of Mulligan joint mobilizations and trunk stabilization exercises versus isometric knee strengthening in the management of knee osteoarthritis: a randomized controlled trial. BMC Sports Sci Med Rehabil. 2024 May 7;16(1):105. doi: 10.1186/s13102-024-00893-7. PMID 38715135